CLINICAL TRIAL: NCT05045664
Title: Early Stage Follicular LymphOma and RadioTherapy PLUS Anti-CD20 Antibody
Acronym: FORTplus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Klaus Herfarth, MD, Vice Chair, Department of Radiation Oncology, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-000362-15
Record Dates: First submitted 2021-08-25; First posted 2021-09-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Early Stage Follicular Lymphoma WHO Grade 1/2 or 3a
MeSH Terms: interventions — Rituximab; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Controlled, open, randomised, 2 parallel groups, multi-centre, national, treatment phase III trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard (Active Comparator): Standard dose (24 Gy) involved site radiotherapy plus Rituximab
  Interventions: Radiation: Standard; Drug: Standard
- Experimental (Experimental): ow-dose (4 Gy) involved site radiotherapy in combination with Obinutuzumab
  Interventions: Radiation: Experimental; Drug: Experimental

INTERVENTIONS:
Radiation: Standard — 12 x 2 Gy involved site radiotherapy plus Rituximab
  Arms: Standard
Radiation: Experimental — 2 x2 Gy involved site radiotherapy plus Obinutuzumab
  Arms: Experimental
Drug: Standard — Rituximab with 12 x 2 Gy involved site radiotherapy
  Other Names: Rituximab
  Arms: Standard
Drug: Experimental — Obinutuzumab with 2 x2 Gy involved site radiotherapy
  Other Names: Obinutuzumab
  Arms: Experimental

SUMMARY:
The MIR study proved the effect of Rituximab in combination with a localized irradiation given in a standard dose. Together with the TROG 99.03 trial, this led to the recommendation of using this combined approach in early stage nodal follicular lymphoma. The GAZAI study is currently looking for the effect of a low dose radiotherapy of 2x2 Gy in combination with Obinutuzumab. The combination seems to show a high CR rate based on the 50% of the patients. This is in contrast to the FORT trial, which showed an inferiority of the 4 Gy dose compared to the standard dose (24 Gy) in terms of response and progression free survival.

The goal of the FORTplus trial is to prove (1) the non-inferiority of LDRT (4Gy) in a combined approach with an anti-CD20-antibody. In case of non-inferiority, a possible (2) superiority of the Obinutuzumab + LDRT should be tested against Rituximab + standard dose using the same test set.

The radiation dose can significantly be reduced to 16% of the standard dose if (1) is confirmed. Knowing the data of the FORT trial, this would have a significant influence on the treatment of the disease worldwide even if the difference in the CR rate at week 18 is not as high as currently in the historical comparison expected.

ELIGIBILITY:
Inclusion Criteria:

* • Centrally reviewed CD20-positive follicular lymphoma grade 1/2 or 3a based on WHO classification (2008)

  * Untreated (radiation-, chemo- or immunotherapy) nodal follicular lymphoma (including involvement of Waldeyer´s ring)
  * Age: ≥18 years
  * ECOG: 0-2
  * Stage: clinical stage I or II (Ann Arbor classification) based on FDG-PET Staging
  * Risk profile: Largest diameter of the lymphoma ≤ 7 cm (sectional images)
  * Written informed consent and willingness to cooperate during the course of the trial
  * Adequate bone marrow capacity: ANC ≥ 1.5 x 103/ml, thrombocytes ≥ 100000 x 10 3/ml, hemoglobin ≥ 10 g/dL
  * Capability to understand the intention and the consequences of the clinical trial
  * Adequate contraception for men and women of child-bearing age during therapy and 18 months thereafter

Exclusion Criteria:

* Extra nodal manifestation of follicular lymphoma
* Secondary cancer in the patient's medical history (exclusion: basalioma, spinalioma, melanoma in situ, bladder cancer T1a, non-metastasized solid tumor in constant remission, which was diagnosed >3 years ago)
* Serious disease interfering with a regular therapy according to the study protocol, e.g: congenital or acquired immune-deficiency syndromes, active infections including viral hepatitis, uncontrolled concomitant diseases including significant cardiovascular or pulmonary disease
* Severe psychiatric disease
* Pregnancy / lactation
* Known hypersensitivity against Obinutuzumab or Rituximab drugs with similar chemical structure or any other additive of the pharmaceutical formula of the study drug
* Active hepatitis B infection (inactive hepatitis B infections require additional prophylactic anti-viral medication for 1 year (e.g. Lamivudin, Entecavir, Tenofovir)
* Participation in another interventional trial or follow-up period of a competing trial which can influence the results of this current trial
* Creatinine > 1.5 times the upper limit of normal (ULN) (unless creatinine clearance normal), or calculated creatinine clearance < 40 mL/min
* AST or ALT > 2.5 × ULN
* Total bilirubin ≥ 1.5 × ULN
* INR > 1.5 × ULN
* PTT or aPTT > 1.5 × the ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Morphologic complete response | Week 18
  Rate of morphologic complete response based on CT scan in patients with initially remaining lymphoma

SECONDARY OUTCOMES:
Metabolic complete response | week 18
  Rate of metabolic complete response based on FDG PET in patients with initially remaining lymphoma
Morphologic response | Month 6
  Morphologic CR in patients with initially remaining lymphoma
PFS | 2 years
  Progression-free survival (PFS) of each treatment arm
Frequency and extent of Toxicity | until month 30
  Toxicity (NCI-CTC criteria, version 5) of all patients
Overall survival | 2 years
  Overall survival (OS) of each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Herfarth, MD, Principal Investigator — Heidelberg University
Locations (12):
- Germany (12):
  - Vivantes Klinikum Berlin, Berlin
  - University of Essen, Essen
  - University of Göttingen, Göttingen
  - University Hospital Heidelberg, Heidelberg
  - Strahlentherapie KH Maria Hilf, Mönchengladbach
  - LMU München, Munich
  - Technische Universität München, Munich
  - Krankenhaus Barmherzige Brüder, Regensburg
  - University of Rostock, Rostock
  - Katharinen Hospital Stuttgart, Stuttgart
  - University of Tübingen, Tübingen
  - University of Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konig L, Dreyling M, Durig J, Engelhard M, Hohloch K, Viardot A, Witzens-Harig M, Kieser M, Klapper W, Pott C, Herfarth K. Therapy of nodal Follicular Lymphoma (WHO grade 1/2) in clinical stage I/II using response adapted Involved Site Radiotherapy in combination with Obinutuzumab (Gazyvaro) - GAZAI Trial (GAZyvaro and response adapted Involved-site Radiotherapy): a study protocol for a single-arm, non-randomized, open, national, multi-center phase II trial. Trials. 2019 Aug 30;20(1):544. doi: 10.1186/s13063-019-3614-y. PMID 31470902
- [Background] Hoskin PJ, Kirkwood AA, Popova B, Smith P, Robinson M, Gallop-Evans E, Coltart S, Illidge T, Madhavan K, Brammer C, Diez P, Jack A, Syndikus I. 4 Gy versus 24 Gy radiotherapy for patients with indolent lymphoma (FORT): a randomised phase 3 non-inferiority trial. Lancet Oncol. 2014 Apr;15(4):457-63. doi: 10.1016/S1470-2045(14)70036-1. Epub 2014 Feb 24. PMID 24572077
- [Result] Herfarth K, Borchmann P, Schnaidt S, Hohloch K, Budach V, Engelhard M, Viardot A, Engenhart-Cabillic R, Keller U, Reinartz G, Eich HT, Witzens-Harig M, Hess CF, Dorken B, Durig J, Wiegel T, Hiddemann W, Hoster E, Pott C, Dreyling M. Rituximab With Involved Field Irradiation for Early-stage Nodal Follicular Lymphoma: Results of the MIR Study. Hemasphere. 2018 Nov 30;2(6):e160. doi: 10.1097/HS9.0000000000000160. eCollection 2018 Dec. PMID 31723798
- [Result] Hoskin P, Popova B, Schofield O, Brammer C, Robinson M, Brunt AM, Madhavan K, Illidge T, Gallop-Evans E, Syndikus I, Clifton-Hadley L, Kirkwood AA. 4 Gy versus 24 Gy radiotherapy for follicular and marginal zone lymphoma (FoRT): long-term follow-up of a multicentre, randomised, phase 3, non-inferiority trial. Lancet Oncol. 2021 Mar;22(3):332-340. doi: 10.1016/S1470-2045(20)30686-0. Epub 2021 Feb 1. PMID 33539729